CLINICAL TRIAL: NCT07012057
Title: A Phase II Open-Label Study of Deucravacitinib for Refractory Adults With Dermatomyositis/ Juvenile Dermatomyositis
Brief Title: Study of Deucravacitinib for Refractory Adults With Dermatomyositis/Juvenile Dermatomyositis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer discontinued investigational drug supply.
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002167; 002167-AR
Record Dates: First submitted 2025-06-07; First posted 2025-06-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Myositis; Dermatomyositis
Keywords: Dermatomyositis; Myositis; Juvenile Dermatomyositis; Deucravacitinib; Janus Kinase Inhibitor
MeSH Terms: conditions — Myositis; Dermatomyositis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug (Deucravacitinb) (Experimental): Participants will receive a 6mg pill taken 2 times per day over 24 weeks and an optional extension period
  Interventions: Drug: Deucravacitinb

INTERVENTIONS:
Drug: Deucravacitinb — Participants will receive a 6mg pill taken 2 times per day over 24 weeks and an optional extension period

SUMMARY:
Background:

Dermatomyositis (DM) and juvenile dermatomyositis (JDM) are diseases that weaken the immune system. DM and JDM can affect the muscles, skin, joints, and lungs and cause skin rashes and muscle inflammation. Symptoms include weakness, pain, fatigue, and rash. Not everyone responds to current treatments. The FDA has approved a drug called deucravacitinib to treat people with plaque psoriasis. Researchers want to find out if this drug can help people with DM or JDM, too.

Objective:

To test deucravacitinib in people with DM or JDM.

Eligibility:

People aged 18 years and older with DM or JDM.

Design:

Participants will have 9 clinic visits over 28 weeks.

Participants will be screened. They will have a physical exam with blood and urine tests. They will have a test of their heart function. They will complete a short questionnaire about their daily life, pain level, and ability to walk, eat, and do other activities.

Deucravacitinib is a pill taken by mouth twice per day at home. Participants will come to the clinic once every 4 weeks for 24 weeks while they are taking the drug. They will have a final visit 4 weeks after their last dose of the study drug. Blood and urine tests will be repeated during these visits. Each visit may take up to 6 hours.

If the drug is helping them, participants may extend their treatment beyond the first 24 weeks. Then they will visit the clinic every 3 months.

DETAILED DESCRIPTION:
Study Description:

Myositis is a heterogeneous family of systemic autoimmune diseases affecting adults and children that can affect the muscle, skin, lungs, joints, and/or gastrointestinal tract. Unfortunately, many patients do not respond completely to current immunosuppressive therapies. Although the pathophysiological mechanisms underlying these diseases are incompletely understood, in adult patients with dermatomyositis (DM) and juvenile dermatomyositis (JDM), a Type 1 interferon gene signature in blood, skin, and muscle correlates with disease activity. Furthermore, recent reports suggest that non-selective inhibitors of the JAK/STAT pathway may be effective in treating patients with refractory DM and JDM. In this study, we will test our hypothesis that inhibition of JAK/STAT pathway using the selective oral TYK2 inhibitor, deucravacitinib, will be efficacious and safe in adult patients with active, treatment-refractory DM/JDM by performing a 24-week, phase II, open-label treatment trial.

At the conclusion of the Treatment Period of the study, all subjects will have the option to receive deucravacitinib in the Extension Portion of the trial.

Objectives:

Primary Objective:

To obtain preliminary data regarding the efficacy of a selective TYK2 inhibitor, deucravacitinib, in adult patients with active, treatment-refractory DM/JDM, as defined by the 2016 ACR/EULAR Criteria for Minimal, Moderate, and Major Clinical Response in Adults with Dermatomyositis and Juvenile Dermatomyositis.

Exploratory Objectives:

* To obtain preliminary data regarding the efficacy of deucravacitinib to improve skin disease activity in adult patients with active, treatment-refractory JDM/DM, as defined by the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI).
* To obtain preliminary data regarding the frequency and incidence of adverse events in treatment-refractory DM/JDM patients treated with deucravacitinib.

Endpoints:

Primary endpoint:

The number of DM/JDM patients achieving at least a "minimal clinical response" using the total improvement score as defined in the 2016 ACR/EULAR Criteria for Minimal, Moderate, and Major Clinical Response in Adult Dermatomyositis and Polymyositis and Juvenile Dermatomyositis at 24 weeks of treatment.

Exploratory endpoints:

* The number of DM/JDM patients with significantly improved skin disease activity (>14 point decrease out of 100) as measured by the CDASI at 24 weeks of treatment.
* The frequency and incidence of treatment-related adverse events reported and observed. (Time Frame: At 28 weeks)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, 18 years of age or older, of any race or ethnicity.
* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to take oral medication and willingness to adhere to the deucravacitinib regimen.
* Definite or probable dermatomyositis or juvenile onset dermatomyositis by ACR/EULAR criteria
* Refractory myositis as defined by intolerance or inadequate response to at least a 12-week trial of corticosteroids and at least one other first line immunomodulatory agent. The definition of intolerance is side effect(s) that require discontinuation of the medication or an underlying condition that precludes the further use of the medication. Adequate treatment with corticosteroids or immunomodulatory drugs is defined as at least the lowest of the following doses:

  * Corticosteroids: 20mg/day for at least 4 weeks with total duration at any dose for at least 12 weeks. If there is intolerance, trial must be for at least 2 weeks.
  * Methotrexate: 15 mg/week for 12 weeks
  * IVIg: 1 g/kg/month or 60 g/month for 3 months
  * Azathioprine: 150 mg/d for at least 12 weeks
  * Mycophenolate mofetil: 1000 mg twice daily for at least 12 weeks
  * Cyclophosphamide: 500 mg/month intravenously for at least 3 months
  * Tacrolimus: 5 mg/d for at least 12 weeks
  * Cyclosporine: 2.4 mg/kg/d for at least 12 weeks
  * Rituximab: 750mg for at least 2 infusions
  * Adalimumab: 40mg SQ every other week for at least 12 weeks
  * Infliximab: 1000mg every 4 weeks for at least 12 weeks
  * Abatacept:

    * IV 10mg/kg or 750mg every 4 weeks for 12 weeks
    * SQ 125mg weekly for at least 12 weeks
  * Tocilizumab:

    ---IV 800mg every 4 weeks for at least 12 weeks
  * SQ 162mg/dose every 2 weeks for at least 12 weeks

Note: Doses/Timelines may be shorter will still qualify if there is documented intolerance. Other medications can be accepted on a case-by-case basis in consultation with the safety committee.

* Concurrent medications: Corticosteroids and non-biologic immunosuppressive/ immunomodulatory drugs can be continued on study. IVIg can also be continued on study. Study participants must be on at least one immunomodulatory medication when enrolling on this study as standard therapy.
* Active disease based on Manual Muscle Testing (MMT-8) of <136/150 and any 1 of the following core disease activity measures:

  1. Physician global activity of >= 3.0/10.0
  2. Patient global activity of >= 3.0/10.0
  3. Extramuscular global activity of >= 3.0/10.0
  4. Health Assessment Questionnaire (HAQ) score of >= 0.75
* Women of child-bearing potential must be willing to undergo pregnancy testing at every on-site visit for the duration of the study.
* For females of reproductive potential: use of highly effective contraception for at least one month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of deucravacitinib administration.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
* Must be English-speaking

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Prior use of a JAK inhibitor.
* Use of other investigational drugs at the time of enrollment.
* Rituximab use within 6 months.
* If rituximab given within 12 months, absence of detectable CD20 cells.
* Concurrent use of any biologic agent other than IVIG.
* Cyclophosphamide use within 12 months.
* Prednisone dose greater than 20 mg/day.
* Change in dose of prednisone within 4 weeks prior to the baseline timepoint.
* Prednisone at a dose of 80 mg or more within 4 weeks prior to baseline timepoint.
* Intravenous methylprednisolone within 8 weeks prior to baseline timepoint.
* Change in dose of methotrexate, azathioprine, mycophenolate, leflunomide, IVIG, cyclosporine, hydroxychloroquine, or tacrolimus within 12 weeks prior to the baseline timepoint.
* History of hypersensitivity to the study drug or drugs of similar chemical classes.
* Late-stage DM patients whose muscle weakness, according to the Investigator, could be attributable to muscle damage rather than myositis disease activity.
* Patients with other types of myositis or myopathies: polymyositis, paraneoplastic myositis, inclusion body myositis, metabolic or drug induced myopathy, dystrophies.
* Patients with history of positive anti-Jo1 or other antisynthetase autoantibodies.
* Patients with advanced clinically symptomatic interstitial lung disease.
* Pregnant or breast-feeding patients.
* History of or active rapidly-progressive interstitial lung disease.
* History of bowel rupture or inflammatory bowel diseases.
* Evidence of latent or active tuberculosis or mycobacterial infections.
* Recent infection requiring antibiotics in the past 4 weeks before entry of study.
* History of any malignancy of any organ system (other than localized basal cell carcinoma of the skin or cutaneous squamous cell carcinoma in situ), treated or untreated, within the past 3 years, regardless of whether there is evidence of local recurrence or metastases.
* Evidence of any other acute or chronic infectious diseases, including hepatitis, HIV, TB, etc.
* Have had symptomatic herpes zoster infection within 12 weeks prior to entry or during the screening period or recurrent herpes simplex infection
* Have a history of disseminated/complicated herpes zoster (for example, multidermatomal involvement, ophthalmic zoster, central nervous system involvement, postherpetic neuralgia)
* Have received any live or live attenuated vaccines (including varicella or measles) within 2 months prior to study enrollment.
* Current or recent history of uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease.
* Any other condition or criterion that, in the judgment of the Investigator, would either pose an unacceptable risk to the participant or interfere with the interpretation of the study results.
* Adults who lack capacity to consent.
* Have a history of chronic alcohol abuse or intravenous drug abuse within the 2 years prior to entry.
* History of previous blood clot such as deep vein thrombosis, pulmonary embolus, or other significant increased risk for blood clots
* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have joint disease or other musculoskeletal condition including contractures or calcinosis, which precludes the ability to quantitate muscle strength.
* Hospitalization within the past 30 days, other than scheduled infusion or procedure.
* Total WBC count <2500 cells/microliter; Absolute neutrophil count <= 1000/mm3; platelets <= 100,000/microliter; hemoglobin <= 10gm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
To obtain preliminary data regarding the efficacy of a selective TYK2 inhibitor, deucravacitinib, in adult patients with active, treatment-refractory DM/JDM | At 24 weeks
  The number of DM/JDM patients at least a minimal Clinical response using the total improvement score as defined in 2016 ACR/EULAR Criteria for Minimal, Moderate, and Major Clinical Response in Adult Dermatomyositis and Polymyositis and Juvenile Dermatomyositis

SECONDARY OUTCOMES:
To obtain preliminary data regarding the efficacy of deucravacitinib to improve skin disease activity in adult patients with active, treatment-refractory DM/JDM, as defined by the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) | At 24 weeks
  The number of DM/JDM patients with significantly improved skin disease (>14 point decrease out of 100) as measured by the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
To obtain preliminary data regarding the frequency and incidence of adverse events in treatment-refractory dermatomyositis patients treated with deucravacitinib. | Over 28 weeks
  The frequency and incidence of treatment-related adverse events reported and observed

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Mammen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002167-AR.html